CLINICAL TRIAL: NCT03115008
Title: Training for COMPLETE Polyp Resection During Colonoscopy -Improving Competency and Metrics for PoLypectomy Skills Using Evaluation Tools and VidEo Feedback
Brief Title: Improving Competency and Metrics for PoLypectomy Skills Using Evaluation Tools and VidEo Feedback (COMPLETE)
Acronym: COMPLETE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: University of Colorado, Denver (Other); Colorado Clinical & Translational Sciences Institute (Other); University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Tonya Kaltenbach, Associate Professor of Clinical Medicine, San Francisco Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: COMPLETE 16-21096
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-based terminal feedback (Experimental)
  Interventions: Behavioral: Video-based terminal feedback
- Conventional concurrent feedback (No Intervention)

INTERVENTIONS:
Behavioral: Video-based terminal feedback — Terminal feedback is given after skill performance using video-based coaching coupled with a validated polypectomy assessment tool
  Arms: Video-based terminal feedback

SUMMARY:
I plan to investigate the value of video-based feedback in endoscopic training - specifically, the role of terminal video feedback as compared to usual concurrent feedback on cold snare polypectomy technique in trainees, using Direct Observation of Polypectomy Skills (DOPyS) competency score. I have focused the study on the competency of cold snare polypectomy for subcentimeter polyps. The majority (>75%) of colon polyps are smaller than one centimeter. Cold snare polypectomy has been shown, and recommended by the American Society for Gastrointestinal Endoscopy (ASGE), to be an effective removal technique. However, its widespread use and moreover, its teaching to trainees is lacking. It takes time and resources to learn and teach endoscopic techniques. Our study will hope to identify a mechanism through video-based feedback that could help to improve the translation of the training of polypectomy skills to its actual performance, and to accelerate the learning curve.

ELIGIBILITY:
Inclusion Criteria:

* Participants: Senior level UCSF gastroenterology trainees (2nd and 3rd year GI fellows) rotating at the San Francisco Veterans Affairs Medical Center (SFVAMC).
* Patients undergoing elective routine colonoscopy procedure.

Exclusion Criteria:

* Participants: Junior level University of California, San Francisco (UCSF) gastroenterology trainees (1st year GI fellows) rotating at the San Francisco Veterans Affairs Medical Center, and senior level trainees who are not rotating at the SFVAMC.
* Patients: Patients undergoing undergoing emergency colonoscopy procedure.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Number of polypectomies for gastroenterology trainees to achieve competency | 2 years
  Observing cold snare polypectomy of polyps <1cm as assessed by DOPyS (score greater or equal to 3)

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States

REFERENCES:
- [Derived] Kaltenbach T, Patel SG, Nguyen-Vu T, Malvar C, Keswani RN, Hall M, Aagaard E, Asokkumar R, Chin YK, Hammad H, Rastogi A, Shergill A, Simon V, Soetikno A, Soetikno R, Wani S. Varied Trainee Competence in Cold Snare Polypectomy: Results of the COMPLETE Randomized Controlled Trial. Am J Gastroenterol. 2023 Oct 1;118(10):1880-1887. doi: 10.14309/ajg.0000000000002368. Epub 2023 Jun 13. PMID 37307537